CLINICAL TRIAL: NCT00001183
Title: Comprehensive Evaluation of the Etiology and Pathogenesis of Chronic Lung Disease (Screening Protocol)
Brief Title: Evaluation of the Causes and Disease Processes of Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 820032; 82-H-0032
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Disease
Keywords: Computed Tomography; Fiberoptic Bronchoscopy; Pulmonary Function Testing; Cardiopulmonary Exercise Testing; Allergen Skin Testing
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Pulmonary Patients

SUMMARY:
Chronic lung diseases are disorders associated with abnormalities in any of the structures involved in the process of breathing and bringing oxygen into the lungs and blood. This includes abnormalities in the airways, lungs, blood vessels in and around the lungs, and the tissue covering the lungs (pleura).

The purpose of this research study is to evaluate patients referred to the Cardiovascular and Pulmonary Branch of the National Heart, Lung, and Blood Institute (NHLBI) in order to;

1. Develop a better understanding of the causes and disease processes involved in disorders of the lungs
2. Identify patients eligible to participate in other P-CCMB research studies

DETAILED DESCRIPTION:
The chronic lung diseases are those disorders associated with functional and/or structural derangement to the alveolar structures, airways, pulmonary blood vessels, pleura and/or mediastinum. The purpose of this project is to permit the comprehensive evaluation of patients referred to the Pulmonary Branch of the National Heart, Lung, and Blood Institute (NHLBI) in order to: (1) develop an understanding of the etiology and pathogenesis of these disorders; and (2) identify individuals who will be suitable candidates for other NHLBI protocols. Testing and procedures will only be performed when medically indicated for the purposes of making a diagnosis or obtaining information likely to be useful in the management of the subjects' disease or condition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Symptoms consistent with pulmonary disease.

May have family history of lung disease.

Patients with diseases of organs with known association with lung disease.

Ranging in age from 7 to 90 years old.

Pregnant and nursing women may participate in minimal risk procedures

EXCLUSION CRITERIA:

Persons with no clinical evidence of lung disease.

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients being screened for lung disease
Sampling Method: Non-Probability Sample
Enrollment: 6564 (Actual)
Dates: Start 1984-11-18 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
N/A-screening protocol | 1 Visit
  Evaluate

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1982-H-0032.html